CLINICAL TRIAL: NCT07302373
Title: Harnessing Endogenous Brain Plasticity Systems for the Recalibration of Pathological Auditory Percepts
Brief Title: Closed-loop Rehabilitation for Hyperactive Hearing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding for this study ended prior to enrollment of any participants.
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Daniel Brandon Polley, Daniel Polley, Professor in Department of Otology and Laryngology, Massachusetts Eye and Ear Infirmary, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: pending_102121
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Tinnitus; Hyperacusis
MeSH Terms: conditions — Tinnitus; Hyperacusis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sound Therapy Group 1 (Experimental): Closed-loop sound therapy. Weekly sessions over 6 weeks.
  Interventions: Behavioral: Sound Therapy 1
- Sound Therapy Group 2 (Placebo Comparator): Placebo sound therapy. Weekly sessions over 6 weeks.
  Interventions: Behavioral: Sound therapy 2

INTERVENTIONS:
Behavioral: Sound Therapy 1 — Closed-loop sound therapy.
  Arms: Sound Therapy Group 1
Behavioral: Sound therapy 2 — Placebo sound therapy.
  Arms: Sound Therapy Group 2

SUMMARY:
There are no widely available treatments for the underserved populations with tinnitus, hyperacusis, and hearing-in-noise deficits. Left unmanaged, these disorders can lead to a wide range of negative psychosocial and emotional sequelae including anxiety, depression, fear, and social isolation. The proposed research will investigate a novel closed-loop sound therapy designed to address the mutual basis of these disorders.

DETAILED DESCRIPTION:
Upwards of 700 million people are projected to require rehabilitative services for hearing disorders by the year 2050 (Chadha, Kamenov, & Cieza, 2021). Many will suffer not from what is inaudible but from the presence of insuppressible sound. Individuals may be overwhelmed by phantom sounds that do not exist external to the auditory system (tinnitus) (Henry, Dennis, & Schechter, 2005). Moderate intensity sounds may have malformed percepts that induce loudness, annoyance, fear, or pain (hyperacusis) (Tyler et al., 2014). Sounds may also appear engulfed by other noises in the environment (Plack, Barker, & Prendergast, 2014). These hearing disorders are co-morbid with one another with roughly 80% of tinnitus patients reporting reduced sound level tolerance (Anari et al., 1999). Hyperacusis, tinnitus, and hearing-in-noise deficits are common chronic disorders within middle-aged/older adults but can also affect younger ages, with noise exposure history and traumatic brain injuries as key predictors. The outlined hearing disorders are complicated and heterogeneous making them challenging to treat. Consequently, despite a clear demand for rehabilitative services, there are no widely accepted nor effective treatments available (Baguley and Hoare, 2018). The result of this is typified in tinnitus patients, of whom 84.8% have never attempted any form of remedy (Bhatt, Lin, & Bhattacharyya, 2016).

We propose a therapeutic strategy that is founded upon the most beneficial aspects of previously conducted randomized controlled trials (RCTs). Namely, the therapy will employ a closed-loop system. The research capitalizes on promising findings from current studies in animal models, seeking to take advantage of the neuroscience principles thought to operationalize paired plasticity. The therapy is entirely non-invasive, posing minimal risk to the patient, and is translatable to widely available hardware. The research will use a "gold-standard" randomized, double-blinded, placebo-controlled clinical trial to objectively evaluate its worth.

ELIGIBILITY:
Inclusion Criteria:

* Normal audiometric thresholds
* Subjects with tinnitus will have self-reported chronic tinnitus that has persisted for the duration of at least 6 months
* Subjects with hyperacusis will have a clinical diagnosis of hyperacusis and/or self-reported sound tolerance complaints that have persisted for the duration of at least 6 months

Exclusion Criteria:

* Conductive hearing loss (as assessed by audiologist)
* Active otologic disease (as assessed by audiologist)
* Significant cognitive decline (Montreal Cognitive Assessment score > 25)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-21 (Estimated); Primary Completion 2023-09-21 (Estimated); Study Completion 2023-09-21 (Estimated)

PRIMARY OUTCOMES:
Change in Score on the Tinnitus Reaction Questionnaire | Pre-test / Post-test (6 weeks) / Follow-up (14 weeks)
Reduction in Loudness Discomfort Levels | Pre-test / Post-test (6 weeks) / Follow-up (14 weeks)
  The intensity of pulsated pure tones of 55 ms reported to be uncomfortably loud (test commonly employed in hearing aid fitting).
Change in Speech Recognition in Noise Performance Accuracy | Pre-test / Post-test (6 weeks) / Follow-up (14 weeks)
  Keyword recognition accuracy for sentences in noise will be assessed with a clinical test, the QuickSiN. Signal to noise ratios vary from 25 to 0 dB in 5 dB steps.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Polley, Ph.D., Principal Investigator — Massachusetts Eye and Ear Infirmary